CLINICAL TRIAL: NCT07321548
Title: Investigating the Gut Microbiota of Individuals With Adenoma, Advanced Adenoma and Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Institute of Gastroenterology and Hepatology, Vietnam (Other); Mahidol University (Other); National University of Malaysia (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jessie Qiaoyi Liang, Research Associate Professor, Chinese University of Hong Kong
Other Study IDs: CREC 2021.036
Record Dates: First submitted 2025-12-18; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Colorectal Adenoma; Colorectal Neoplasms
Keywords: Gut Microbiome; Non-invasive Test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples collected from subjects and the derivatives will be retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- N: Healthy control
  Interventions: Diagnostic Test: Fecal immunochemical test
- nAA: Subject diagnosed with non-advanced adenoma
  Interventions: Diagnostic Test: Fecal immunochemical test
- AA: Subject diagnosed with advanced adenoma
  Interventions: Diagnostic Test: Fecal immunochemical test
- CRC: Subject diagnosed with colorectal cancer
  Interventions: Diagnostic Test: Fecal immunochemical test

INTERVENTIONS:
Diagnostic Test: Fecal immunochemical test — This diagnosis test is commonly used for screening CRC, which can act as an indicator to compare the performance of our new molecular test

SUMMARY:
This observational study aims to help establish the first molecular test for non-invasive prediction of recurrent adenoma, which will help identify patients at high risk of recurrent adenoma for further colonoscopy examination, and validate the microbial test for CRC screening in different populations.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignancies worldwide. CRC is now the commonest cancer and the second cause of cancer death in Hong Kong. Most CRCs begin as small polyps. Some polyps in particular adenomas may gradually develop into cancer. Early detection of cancer can facilitate successful treatment, and early detection of adenomas can prevent and decrease CRC incidence. Therefore, many efforts are being made to screening of colorectal adenoma and cancer, which will benefit public health greatly in Hong Kong and worldwide.

Abnormality in the composition of the gut microbiota has been implicated as a potentially important etiological factor in the initiation and progression of CRC. With the widespread application of metagenomic analyses in the investigation of intestinal microbiota, an increasing number of bacteria have been identified to be positively associated with CRC. Recent basic research has established a critical function for the intestinal microbiota and specific bacterial species, in promoting colorectal tumorigenesis.

Based on the previously identified microbial markers, the investigators have recently proven that fecal microbial markers can also serve in non-invasive diagnosis of recurrent adenoma in post polypectomy patients. The results have shown that, the panel of microbial markers composing of Fusobacterium nucleatum (Fn), Bacteroides clarus (Bc), Clostridium hathewayi (Ch), and the Lachnoclostridium marker m3 shows good diagnostic performance for colorectal adenoma and CRC. Microbial markers can be used to predict risk of adenoma recurrence during follow-up surveillance, with different scoring algorithms and cutoff values as compared to those used for colorectal neoplasm screening. However, only retrospective samples were used in the previous study, and sample size was limited. A prospective study is warranted to verify the accuracy of the microbial test for predicting recurrent adenoma.

ELIGIBILITY:
Inclusion Criteria:

* History of polypectomy or surgical removal of adenoma or CRC within the past 10 years
* Will undergo a scheduled standard colonoscopy examination

Exclusion Criteria:

* History of inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population scheduled for colonoscopy of participating country/city will be invited and recruited in wards, clinics or endoscopy centres.
Sampling Method: Non-Probability Sample
Enrollment: 1757 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Determine the performance of microbial markers in predicting adenoma and CRC | 3 months after stool sample submission

SECONDARY OUTCOMES:
Compare microbiome composition between healthy subjects and populations with adenoma, advanced adenoma, and colorectal cancer | Approximately 1 year after completed subject recruitment of the study
Delineate the gut microbial community profiles of the population with adenoma, advanced adenoma, and colorectal cancer residing in different geographical locations with different lifestyles | Approximately 1 year after completed subject recruitment of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No